CLINICAL TRIAL: NCT05437991
Title: Ultrasonographic Morphology Assessment of Low-grade Carotid Stenosis
Acronym: QUAMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-CHITS-005; 2022-A00854-39 (Other: ID-RCB)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-10

CONDITIONS: Carotid Stenosis
Keywords: Low-grade carotid stenosis; Ultrasound imaging; Morphological quantification; European Carotid Surgical Trial (ECST); North American Symptomatic Carotid Endarterectomy Trial (NASCET)
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morphological quantification of low-grade carotid stenosis (Other): Morphological quantification using ECST method and implying two independent observers
  Interventions: Diagnostic Test: Independent morphological quantifications by echo-doppler using ECST method

INTERVENTIONS:
Diagnostic Test: Independent morphological quantifications by echo-doppler using ECST method — The physician who is usually in charge of patient follow-up performs a first evaluation of carotid stenosis percentage by echo-doppler using ECST method. Then a second physician immediately performs a second evaluation using the same echo-doppler device without knowing first evaluation conclusions.

SUMMARY:
Internal carotid artery (ICA) is intended to supply blood to brain. The carotid bulb located upstream of ICA origin is prone to atherosclerosis. This is an accumulation of fat and calcium in the wall forming a plaque that gradually thickens and leads to carotid stenosis (CS), which causes a decrease in blood flow. The risk of CS is stroke caused either by carotid artery thrombosis (occlusion) or by atherosclerotic plaque fragmentation, some components of which may leak into the brain (embolism).

When diagnosing CS, an Echo-Doppler is performed to determine bulb and ICA origin obstruction rates. The reference method of quantifying CS is based on hemodynamic criteria that only allow the diagnosis of high grade stenosis thresholds (50%-70%). Below 50%, low-grade stenosis, patient follow-up is limited and could be based on morphological criteria; ultrasound imaging being a reference technique for human body structures morphological assessment, especially vessels.

Two methods of CS morphological quantification with Doppler ultrasound currently exist. Calibre reduction at the maximum of stenosis can be measured by relating the smallest luminal diameter to the vessel diameter at stenosis site (ECST method) or to the downstream ICA diameter (NASCET method). As bulb diameter measures ≈1.8 times that of ICA, ECST appears to be more suitable for CS quantification. For high-grade stenosis, morphological quantification performance is impaired due to extensive calcification of large atheromatous plaques. However, it is possible that less calcified nature of low-grade stenosis and the use of a rigorous methodology will allow reproducible assessment in routine practice. This technique has not yet been evaluated, although it is a frequent situation in patient follow-up.

DETAILED DESCRIPTION:
Internal carotid artery is intended to supply blood to brain. The carotid bulb located upstream of internal carotid artery origin is prone to atherosclerosis. This is an accumulation of fat and calcium in the wall, forming a plaque which gradually thickens and leads to carotid stenosis, causing a reduction in blood flow. The risk of carotid stenosis is stroke caused either by carotid artery thrombosis (occlusion) or by atherosclerotic plaque fragmentation, some components of which may leak into the brain (embolism).

When carotid stenosis is diagnosed, an Echo-Doppler is performed to determine the bulb and internal carotid artery origin obstruction rates. The reference method for quantifying carotid stenosis is based on hemodynamic criteria that only allow the diagnosis of high grade stenosis thresholds (50%-70%). Below 50%, low-grade stenosis, patient follow-up is limited and could be based on morphological criteria; ultrasound imaging being a reference technique for human body structures morphological assessment, especially vessels.

Two methods of carotid stenosis morphological quantification with Doppler ultrasound currently exist. Calibre reduction at the maximum of stenosis can be measured by relating the smallest luminal diameter to the vessel diameter at stenosis site ("European Carotid Surgical Trial" (ECST), European method) or to the downstream internal carotid artery diameter ("North American Symptomatic Carotid Endarterectomy Trial" (NASCET), North American method). As bulb diameter measures ≈1.8 times that of the internal carotid artery, the NASCET appears to be more suitable for carotid stenosis quantification. For high-grade stenosis, morphological quantification performance is impaired due to extensive calcification of large atheromatous plaques. However, it is possible that less calcified nature of low-grade stenosis and the use of a rigorous methodology will allow reproducible assessment in routine practice.

This technique has not yet been evaluated although it is a frequent situation in patient follow-up. This study therefore suggests to evaluate the inter-observer reproducibility of morphological quantification of these stenosis by the ECST method with a precise methodology.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient referred for Echo-Doppler exploration of the neck vessels
* Patient 18 years of age or older
* Atheromatous arterial disease with stenosis < 50% (maximum systolic velocity < 125 cm/sec for an angle of 50-60°) in at least one carotid artery

Exclusion Criteria:

* Patient refusal
* Unavailability of two physicians to perform examination
* Patient under judicial protection (guardianship, curators...) or justice safeguard
* Pregnant, parturient or breastfeeding woman
* Any other reason that could interfere with study objectives evaluation in the investigator opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the inter-observer reproducibility of morphological quantification of low-grade carotid stenosis (<50%) using the ECST method | 1 day
  Each operators will perform stenosis percentage calculation according to ECST method. Between the two calculations performed independently by the two observers, a difference of ±10% will be considered acceptable.

SECONDARY OUTCOMES:
To assess the performance of morphological quantification technique according to examination feasibility (good, medium, poor). | 1 day
  The examination feasibility will be based on subjective assessment of the conditions under which the measurements are made (systolic and diastolic velocities in the internal carotid artery, diameter of the patent lumen, diameter of the vessel at the site of stenosis):
  * Good: no doubt about measurements accuracy
  * Medium: more difficult to make accurate measurements
  * Poor: significant doubt about measurements accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GIAUFFRET, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Hôpital Sainte Musse, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giauffret F, Hocq F, Lafond S, Autret A, Elias A, European Carotid Surgical Trial-based diameter measurement using B-mode ultrasound imaging to quantify low-grade carotid artery stenosis: the QUAMUS study. JVS-Vascular Insights. Volume 2, 2024, 100061